CLINICAL TRIAL: NCT00139321
Title: Biomechanical Parameters of Gait in Patients With Parkinson's Disease and Parkinsonian Syndromes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Marie-laure Welter, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBM0260
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Gait Disorders, Neurologic
Keywords: Gait disorders; Postural instability; parkinsonian syndrome; Gait initiation; Parkinson's disease; Adults
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation; Parkinsonian Disorders; Parkinson Disease | interventions — Electromyography

INTERVENTIONS:
Device: Force platform and electromyography

SUMMARY:
Gait disorders and falls are frequent in patients with parkinsonian syndromes. In patients with Parkinson's disease (PD), these signs occurred later during the course of the disease in comparison to patients with other degenerative parkinsonian disorders. The pathophysiology of these symptoms are still not fully understood. Gait initiation challenges the balance control system as the body moves from an upright stable static posture to a continuously unstable gait. The aim of this study is to analyse the gait initiation process in patients with parkinsonian disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to walk without assistance
* Patients with Parkinson's disease or other degenerative parkinsonian syndromes (progressive supranuclear palsy [PSP], multiple system atrophy [MSA], corticobasal degeneration [CBD], etc.)

Exclusion Criteria:

* Other parkinsonian syndromes
* Dementia
* Neuroleptic treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Biomechanical gait initiation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yves Agid, MD, PhD, Study Director — CIC-Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France